CLINICAL TRIAL: NCT06495658
Title: The Clinical and Microbial Impact of Prebiotics in Ulcerative Colitis
Brief Title: Impact of Prebiotics in Ulcerative Colitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Berkeley Limketkai, MD, PhD, Associate Clinical Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 24-000256
Record Dates: First submitted 2024-04-03; First posted 2024-07-11 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2024-07

CONDITIONS: Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative | interventions — Prebiotics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and outcomes assessor will not be aware of participants' assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prebiotic at Week 0 (Experimental)
  Interventions: Dietary Supplement: Prebiotic
- Prebiotic at Week 8 (Active Comparator)
  Interventions: Dietary Supplement: Prebiotic

INTERVENTIONS:
Dietary Supplement: Prebiotic — Participants will be asked to take a daily dose of prebiotic supplement for 8 weeks.

SUMMARY:
The cause of inflammatory bowel disease (IBD) is currently unknown, although partly attributed to interactions among genetic risk polymorphisms, environmental factors, gut microbiome, and host immunity. Diet, particularly those with plant-based products, have been shown in prior research to improve gut microbial composition, which has been linked to different IBD-related outcomes. This study is interested in evaluating the impact of prebiotics on gut microbiome composition and gut health in patients with IBD.

Dietary composition will be assessed at baseline and over the course of 16 weeks. Participants will be randomized to either consume an 8-week course of prebiotic supplementation beginning at week 0 or week 8. Stool samples will be collected at weeks 0 and 8. The stool will be analyzed for cross-sectional and longitudinal fecal microbial changes associated with different prebiotic and diet consumption patterns in the context of heterogeneous disease characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 85 years old
* History of biopsy-proven ulcerative colitis (UC)
* Active symptoms (SCCAI >2)
* Concomitant use of 5-aminosalicylates, immunomodulators, and corticosteroids will be permitted, although initiation or dose adjustment must not have occurred within 30 days prior to enrollment.
* Concomitant use of biologic therapy will be permitted, although initiation or dose adjustment must not have occurred within 60 days prior to enrollment.
* Prior probiotics or other dietary supplements use is permitted but will be asked to be discontinued during the course of the trial

Exclusion Criteria:

* Prior colectomy
* Hospitalization
* Urgent need for abdominal surgery
* Unstable major medical condition
* Active malignancy under treatment
* Active alcohol or non-cannabinoid substance abuse
* Pregnancy or lactation
* Concerns for non-compliance

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical response | Week 8
  Clinical response will be defined as a reduction of Simple Colitis Clinical Activity Index (SCCAI). Range of SCCAI is 0-20 (higher is more severe).
Microbial composition | Week 8
  Microbial composition includes a measurement and characterization of the relative quantity of genera and species.

SECONDARY OUTCOMES:
Clinical remission | Week 8
  Clinical remission will be defined as a Simple Colitis Clinical Activity Index (SCCAI) < 4. Range of SCCAI is 0-20 (higher is more severe).
Clinical response | Week 16
  Clinical response will be defined as a reduction of Simple Colitis Clinical Activity Index (SCCAI). Range of SCCAI is 0-20 (higher is more severe).
Clinical remission | Week 16
  Clinical remission will be defined as a Simple Colitis Clinical Activity Index (SCCAI) < 4. Range of SCCAI is 0-20 (higher is more severe).
Microbial composition | Week 16
  Microbial composition includes a measurement and characterization of the relative quantity of genera and species.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No